CLINICAL TRIAL: NCT00001231
Title: The Evaluation of Women With Perimenopause-Related Mood and Behavioral Disorders
Brief Title: Perimenopause-Related Mood and Behavioral Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 880131; 88-M-0131
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-08-18

CONDITIONS: Mood Disorder
Keywords: Mood; Behavior; Cognition; Midlife; Depression
MeSH Terms: conditions — Mood Disorders; Behavior; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Women: The purpose of this protocol is to allow for the careful screening of healthy volunteers for participation in research protocols.
- premenopausal depressed women patients: The purpose of this protocol is to allow for the careful screening of patients for participation in research protocols.

SUMMARY:
The purpose of this study is to investigate mood and behavior changes in the time period surrounding and including menopause. This is an observational study; volunteers who participate will not receive any new or experimental therapies.

Controversy exists regarding the relationship between estrogen and progesterone (gonadal steroid) changes and midlife-onset depression. This study will examine the role of gonadal steroids in perimenopausal mood and behavioral disorders.

Perimenopausal women with depression symptoms and a control group of healthy perimenopausal volunteers will be compared to identify correlates of the occurrence of depression. Participants with depressive symptoms may also participate in companion studies that will test the antidepressant efficacy of phytoestrogens and selective estrogen receptor modulators (SERMS).

A group of younger pre-perimenopausal women with normal menstrual cycle functioning will be followed through menopause in an effort to confirm the association of depression onset with changes in reproductive endocrine functioning....

DETAILED DESCRIPTION:
Controversy exists regarding the relevance of changes in gonadal steroids for midlife onset depressions. The purpose of this protocol is to allow for the careful screening of patients and healthy volunteers for participation in research protocols that examine the role of gonadal steroids in depressions occurring during the perimenopause and for the collection of natural history data. Women in this protocol will undergo an evaluation which may include: a psychiatric diagnostic interview; rating scales; a medical history; a physical exam; blood and urine laboratory evaluation; and a request for medical records. The data collected may also be linked with data from other perimenopausal depression protocols (e.g., DNA, psychophysiology tests, treatment studies, etc.) for the purposes of better understanding the diagnosis, pathophysiology, and treatment response of women with depression during the perimenopause.Upon conclusion of the screening process, participants will either be offered entry into a research protocol and will sign the appropriate informed consent, or will be considered not appropriate for participation in research and will be referred back into the community. The second purpose of this protocol is to permit the identification of premenopausal women who are followed longitudinally through the menopause transition in an effort to confirm the association of depression onset with change in reproductive endocrine function. This protocol, then, serves as a screening and evaluation protocol to recruit subjects who are characterized with standard measures in this protocol and then offered participation in related studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Perimenopausal Subjects:

  * History within the last one year of at least one month with perimenopause-related mood or behavioral disturbances of at least moderate severity - that is, disturbances that are distinct in appearance and associated with a notable degree of functional impairment;
  * Age 40-65;
  * History of the onset of menstrual irregularity during the past six months but not greater than one year of amenorrhea (i.e., not postmenopausal);
  * Biological evidence of a deterioration of normal ovarian activity, specifically, plasma FSH levels persistently elevated (> 14IU/L) (as recommended by the Stages of Reproductive Aging Workshop criteria (106)) drawn at two week intervals over a period of eight weeks;
  * No prior estrogen replacement therapy for treatment of perimenopausal physical or emotional symptoms within the last six months; and
  * In good medical health;
  * Subjects must be competent to comprehend the purpose of the screening process and to provide written informed consent and be willing to participate in NIMH IRB approved research protocols.
* A control group of age-matched perimenopausal women who meet patient selection criteria with the exception of the presence of mood or behavioral disorders will also be sought.
* Premenopausal women will be women who meet the following inclusion criteria for the longitudinal study participants:

  * Regular menstrual cycle function (21-34 days);
  * Absence of current mood or behavioral disturbance as determined by a structured diagnostic interview;
  * Plasma gonadotropin levels in pre-perimenopausal range (<14 IU/L);
  * In good medical health; and
  * Medication free.

EXCLUSION CRITERIA:

* Primary general medical illness (i.e., appears to be causing the mood disorder);
* Current antidepressant therapy (since this is a screening protocol for subsequent treatment studies in which participants must be untreated). Antidepressants will not be withheld from participants who need or want them;
* Current alcohol or substance abuse or dependence (excluding nicotine) of sufficient magnitude to require independent, concurrent treatment intervention (e.g., antabuse or opiate treatment, but not including self-help groups);
* Pregnant or lactating women;
* Subjects who are unable to provide informed consent.
* NIMH employees, staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both depressed and asymptomatic women who are in the perimenopause.
Sampling Method: Non-Probability Sample
Enrollment: 1158 (Actual)
Dates: Start 1989-03-06 (Actual)

PRIMARY OUTCOMES:
Standardized cross-sectional rating scales (Beck Depression Inventory, Hamilton Depression and Anxiety Scales, and the Center for Epidemiologic Studies-Depression Scale), symptom rating scales completed daily, and plasma hormone measures (includ... | Ongoing
  Standardized cross-sectional rating scales (Beck Depression Inventory, Hamilton Depression and Anxiety Scales, and the Center for Epidemiologic Studies-Depression Scale), symptom rating scales completed daily, and plasma hormone measures (including neurosteroid levels).

SECONDARY OUTCOMES:
Plasma ACTH and cortisol response to the o-CRH stimulation tests, selected variants in genomic profile (e.g., SNPs) and genome/exome sequencing, and the results of the SCID interviews | Ongoing
  Plasma ACTH and cortisol response to the o-CRH stimulation tests, selected variants in genomic profile (e.g., SNPs) and genome/exome sequencing, and the results of the SCID interviews

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with dbGaP, BTRIS and NIMH Data Archive as determined by the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 24 months after final publication
Access Criteria: Data will be shared with dbGaP, BTRIS and NIMH Data Archive as determined by the Principal Investigator.

REFERENCES:
- [Background] Kessler RC, McGonagle KA, Swartz M, Blazer DG, Nelson CB. Sex and depression in the National Comorbidity Survey. I: Lifetime prevalence, chronicity and recurrence. J Affect Disord. 1993 Oct-Nov;29(2-3):85-96. doi: 10.1016/0165-0327(93)90026-g. PMID 8300981
- [Background] Schmidt PJ, Rubinow DR. Menopause-related affective disorders: a justification for further study. Am J Psychiatry. 1991 Jul;148(7):844-52. doi: 10.1176/ajp.148.7.844. PMID 2053622
- [Background] Schmidt PJ, Nieman L, Danaceau MA, Tobin MB, Roca CA, Murphy JH, Rubinow DR. Estrogen replacement in perimenopause-related depression: a preliminary report. Am J Obstet Gynecol. 2000 Aug;183(2):414-20. doi: 10.1067/mob.2000.106004. PMID 10942479
- [Derived] Guerrieri GM, Ben Dor R, Li X, Wei SM, Martinez PE, Neiman LK, Rubinow DR, Schmidt PJ. The Cortisol and ACTH Response to Dex/CRH Testing in Women With and Without Perimenopausal Depression. J Clin Endocrinol Metab. 2021 Sep 27;106(10):3007-3018. doi: 10.1210/clinem/dgab407. PMID 34097071
- [Derived] Rudzinskas S, Hoffman JF, Martinez P, Rubinow DR, Schmidt PJ, Goldman D. In vitro model of perimenopausal depression implicates steroid metabolic and proinflammatory genes. Mol Psychiatry. 2021 Jul;26(7):3266-3276. doi: 10.1038/s41380-020-00860-x. Epub 2020 Aug 12. PMID 32788687
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1988-M-0131.html